CLINICAL TRIAL: NCT02908711
Title: Analgesic Efficacy of Adductor Canal Block (ACB) Before and After Primary Total Knee Arthroplasty (TKA): A Prospective Randomized Trial to Compare Postoperative Clinical Outcomes
Brief Title: Adductor Canal Block (ACB) Before and After Primary Total Knee Arthroplasty (TKA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0524-16-RMC
Record Dates: First submitted 2016-08-21; First posted 2016-09-21 (Estimated); Last update posted 2018-09-04 (Actual); Status verified 2016-08

CONDITIONS: Anesthesia, Regional
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients receiving ACB before primary TKA (Active Comparator): Patients receiving adductor canal block (ACB) before primary total knee arthroplasty (TKA).
  Patients randomized to this group will receive the block prior to incision after induction of general anesthesia
  Interventions: Drug: 0.5% ropivacaine
- Patients receiving ACB after primary TKA (Active Comparator): Patients receiving adductor canal block (ACB) immediately after primary total knee arthroplasty (TKA).
  Patients randomized to this group will receive the block at the end of the surgery.
  Interventions: Drug: 0.5% ropivacaine

INTERVENTIONS:
Drug: 0.5% ropivacaine — Adductor canal block (ACB) performed as part of their analgesic regimen for primary total knee arthroplasty achieved with 20 cc of 0.5% ropivacaine under constant ultrasound visualization.

SUMMARY:
Total knee arthroplasty (TKA) is associated with severe postoperative pain. Multimodal analgesia, including peripheral nerve block, is recommended for post-operative pain relief 1. Perineural analgesia offers the advantage of extended pain relief up to 24 hours after surgery2.

This is a prospective, randomized control trial designed to compare the analgesic efficacy of the adductor canal block (ACB) performed immediately before or immediately after primary total knee arthroplasty (TKA). The primary objective of this study is to measure pain score associated with knee motion following TKA among patients receiving ACB as part of their analgesic regimen for TKA. Secondary end points include assessment of postoperative ambulation, range of motion, pain at rest, opioid consumption, and patient satisfaction between the two analgesic approaches. The investigators hypothesize that ACB before the surgery will reduce a patient's postoperative pain and improve patient satisfaction.

All consecutive patients undergoing primary TKA will be recruited for enrollment in the study. Patients will be for randomized preoperatively to receive either preemptive ABC (PreACB) or postoperative ABC (PostACB). Patients randomized to the PreACB group will receive the block prior to incision. Patients randomized to the PostACB group will receive the block at the end of the surgery. Both techniques are in accordance to the standard of care at our institute. All patients will have the ACB done by a regional anesthesiologist in the regional anesthesia unit, or in the operating room. Patient medical history will be obtained and blocks will be placed per usual protocol. Operative and anesthetic details, including medications given, will be recorded.

Pain scores and pain medications given in the PACU will be recorded. Supplementary analgesics will be provided per institutional PACU protocol. Study data will be recorded for up to 72 hours or until patient discharge. A follow-up will occur in 4- 6 weeks at the orthopedic follow-up appointment to evaluate the patient's late pain scores and overall satisfaction. Data will be analyzed both at the conclusion of the study and at several intervals prior to completion of the study.

DETAILED DESCRIPTION:
D. Research Design and Methods

Inclusion Criteria:

The study is a prospective, randomized controlled clinical trial comparing two methods of regional analgesia for primary TKA. All adult primary TKA patients are eligible for inclusion in the study.

Exclusion criteria:

* Allergy to local anesthetics or to systemic opioids
* Contraindication to regional anesthesia technique, such as local infection or coagulopathy
* Sensory/motor disorder involving operative limb
* Requirements of more than 30 mg morphine equivalent daily prior to surgery
* ASA 4 or greater
* Psychiatric or cognitive disorders
* Incarceration
* Renal insufficiency with Cr > 2.0
* Hepatic failure
* Pregnancy
* Age under 18 years Potential risks for the procedure, which will be explained to the patient, include: bleeding, local infection, local anesthetic toxicity. All are commonly listed as rare complications of the procedures.

After consenting to participation and upon randomization, ACBs will be placed either in the regional anesthesia bay or the OR prior to anesthesia induction and surgery, or in the OR immediately upon completion of surgery.

For participating patients, the following data will be collected by the research staff: ASA physical status, age, height, weight, gender, intra- and post operative quantitative opiate use (expressed as morphine equivalent), numeric VAS scores, KSS score (form included) and QoR score (form included).

Those collecting data will be blinded from randomization of patients to either research group.

Intraoperative care:

Intraoperative anesthesia will be achieved using a general anesthetic technique. Intraoperative analgesia will be administered per anesthesiologists' discretion.

All patients will have cemented total knee utilizing a medial parapatellar approach, including patellar resurfacing. A tourniquet will be used in all cases. Posterior capsule infiltration will be done with 20cc of 0.25% bupivacaine, as the preferred method of providing sacral plexus analgesia 5-6, per current institutional protocol.

ACB Procedure Details Patients will lie in the supine position. The needle insertion site, approximately 10cm proximal to their operative knee, will be exposed. The skin will be disinfected with 2% Chlorhexidine and the ultrasound probe placed in a sterile sleeve. The femoral artery is identified with a high frequency linear transducer (Philips 4-12L linear transducer with a frequency of 6-12 MHz, Milwaukee, WI or ) proximal to the operative knee. The appropriate location for injection will be determined by following the femoral artery cephalad until the artery is directly posterior to the Sartorius muscle. At this level, the saphenous nerve is located lateral to the femoral artery. An 18g insulated sonographic Tuohy needle (Pajunk GmbH, Geisingen, Germany) will be inserted in an in-plane approach, under constant ultrasound visualization, through the Sartorius muscle to a final location in close proximity to the saphenous nerve. Once satisfied with needle placement and following negative aspiration, 20 cc of 0.5% ropivacaine will be injected gradually through the needle under visualization, with recurrent aspirations to verify absence of intra-vascular injection signs.

Data Collection Patients will be enrolled for the study during the orthopedic surgical appointment upon the scheduling of the surgery. Upon enrollment, patients will complete a baseline KSS questionnaire (attached), have a VAS pain score recorded, and have their pre-operative analgesic medication documented.

To assess the effect of pain with movement and overall strength, on POD 1, the patient will indicate their level of pain using VAS numeric scale (1-10). QoR questionnaire (attached) will be assessed 24 hours from the placement of the ACB. Overall analgesic medication consumption, both opioid (expressed as morphine equivalent) and non-opioid will be recorded for PODs 1-3.

The patients will also complete the KSS and the QoR questionnaires at the 4-6 week orthopedic follow-up appointment, as VAS scores and total analgesic medication will be documented.

ELIGIBILITY:
Inclusion Criteria:

The study is a prospective, randomized controlled clinical trial comparing two methods of regional analgesia for primary TKA. All adult primary TKA patients are eligible for inclusion in the study.

Exclusion Criteria:

* Allergy to local anesthetics or to systemic opioids
* Contraindication to regional anesthesia technique, such as local infection or coagulopathy
* Sensory/motor disorder involving operative limb
* Requirements of more than 30 mg morphine equivalent daily prior to surgery
* ASA 4 or greater
* Psychiatric or cognitive disorders
* Incarceration
* Renal insufficiency with Cr > 2.0
* Hepatic failure
* Pregnancy
* Age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Pain score associated with knee motion following TKA | 4-6 Weeks postoperatively
  This study's primary endpoint the change in the patient's reported pain score on the preoperative visit, on postoperative day (POD) 1, and the patient's pain score reported on the 4-6 week follow- up visit. Pain score will be measured using a numeric verbal analogue scale (1-10). Pain will be measured using this scale on the pre-operative visit, and on POD1 prior to manipulation, with active (patient driven) movement and with passive (physician elicited) movement.

SECONDARY OUTCOMES:
Opioid consumption | 4-6 weeks postoperatively
  This study secondary endpoints is to evaluate changes in opioid consumption throughout 24-48 hours postoperatively to the 4-6 weeks postoperatively.Opioid consumption will be documented by a member of the research team at 24 hours postoperatively, 48 hours postoperatively , and on the follow-up visit (4-6 weeks postoperatively) in order to identify reduction / increases in patient's opioid consumption trends.
Patient satisfaction between the two analgesic approaches. | 24 hours postoperatively
  Additional secondary endpoint of this study is to evaluate whether patient's satisfaction scores differ amongst the two analgesic approaches on the POD 1. Patient's satisfaction score will be measured using the Quality of Recovery (QoR) score, documented on POD 1.
Assessment of postoperative ambulation. | 4-6 weeks postoperatively
  Additional secondary endpoint of this study include assessment of changes in ambulation the range of motion throughout the study participation, from the preoperative visit to the follow-up visit (4-6 weeks following surgery). Knee Society Score (KSS) will be documented on preoperative visit, on POD 1 and at the follow-up visit ( 4-6 weeks after surgery), to examine changes in ambulation.
Assessment of postoperative pain at rest | 4-6 weeks postoperatively
  Additional secondary endpoint of this study include assessment of changes in pain at rest using the KSS score throughout the study participation, from the preoperative visit to the follow-up visit (4-6 weeks following surgery). Knee Society Score (KSS) will be documented on preoperative visit, on POD 1 and at the follow-up visit ( 4-6 weeks after surgery), to examine changes in patients reported pain at rest.
Thrombo-embolic complications | Up to 24 weeks
  Complications of deep venous thrombosis, pulmonary embolus will be documented
Blood transfusion | Up to 24 weeks
  Additional secondary endpoint of this study is to assess whether the different analgesic approaches effect bleeding complications, measured by the number of patients who receive transfusion of concentrated blood cells units throughout their hospital admission.
Non opioid analgesia consumption | 4-6 weeks postoperatively
  This study secondary endpoints is to evaluate changes in non-opioid analgesia -non opioid medication consumption throughout 24-48 hours postoperatively to the 4-6 weeks after surgery. Non-opioid analgesia - non-opioid medication consumption will be recorded on pre-operative visit, on POD 1, and on the follow-up visit (4-6 weeks postoperatively) in order to identify reduction / increases in patient's non-opioid analgesia -non opioid medication consumption trends.
Patient satisfaction with the two analgesic approaches 4-6 weeks postopertively | 4-6 weeks postoperatively
  Additional secondary endpoint of this study is to evaluate whether patient's satisfaction scores differ among the two analgesic approaches at the follow-up visit (4-6 weeks postoperatively). Patient's satisfaction score will be measured using the Quality of Recovery (QoR) score, documented on follow-up visit.
Abnormal hemoglobin concentration values | Up to 24 weeks
  Additional secondary endpoint of this study is to assess whether the different analgesic approaches effect bleeding complications, measured by the percent of decline in patients' hemoglobin concentration throughout their hospital admission.
Duration of hospital stay | Up to 24 weeks
  Additional secondary endpoint of this study is to assess whether the different analgesic approaches effect duration of hospital admission, measured by the length of stay in the hospital.

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center, Petach Tikvah, Israel

REFERENCES:
- [Background] Fischer HB, Simanski CJ, Sharp C, Bonnet F, Camu F, Neugebauer EA, Rawal N, Joshi GP, Schug SA, Kehlet H; PROSPECT Working Group. A procedure-specific systematic review and consensus recommendations for postoperative analgesia following total knee arthroplasty. Anaesthesia. 2008 Oct;63(10):1105-23. doi: 10.1111/j.1365-2044.2008.05565.x. Epub 2008 Jul 10. PMID 18627367
- [Background] O'Donnell BD, Iohom G. Regional anesthesia techniques for ambulatory orthopedic surgery. Curr Opin Anaesthesiol. 2008 Dec;21(6):723-8. doi: 10.1097/aco.0b013e328314b665. PMID 19009687
- [Background] Jenstrup MT, Jaeger P, Lund J, Fomsgaard JS, Bache S, Mathiesen O, Larsen TK, Dahl JB. Effects of adductor-canal-blockade on pain and ambulation after total knee arthroplasty: a randomized study. Acta Anaesthesiol Scand. 2012 Mar;56(3):357-64. doi: 10.1111/j.1399-6576.2011.02621.x. Epub 2012 Jan 4. PMID 22221014
- [Background] Kang H, Ha YC, Kim JY, Woo YC, Lee JS, Jang EC. Effectiveness of multimodal pain management after bipolar hemiarthroplasty for hip fracture: a randomized, controlled study. J Bone Joint Surg Am. 2013 Feb 20;95(4):291-6. doi: 10.2106/JBJS.K.01708. PMID 23302898
- [Background] Kazak Bengisun Z, Aysu Salviz E, Darcin K, Suer H, Ates Y. Intraarticular levobupivacaine or bupivacaine administration decreases pain scores and provides a better recovery after total knee arthroplasty. J Anesth. 2010 Oct;24(5):694-9. doi: 10.1007/s00540-010-0970-x. Epub 2010 Jun 23. PMID 20571832
- [Background] Essving P, Axelsson K, Aberg E, Spannar H, Gupta A, Lundin A. Local infiltration analgesia versus intrathecal morphine for postoperative pain management after total knee arthroplasty: a randomized controlled trial. Anesth Analg. 2011 Oct;113(4):926-33. doi: 10.1213/ANE.0b013e3182288deb. Epub 2011 Aug 4. PMID 21821506
- [Background] Myles PS, Hunt JO, Nightingale CE, Fletcher H, Beh T, Tanil D, Nagy A, Rubinstein A, Ponsford JL. Development and psychometric testing of a quality of recovery score after general anesthesia and surgery in adults. Anesth Analg. 1999 Jan;88(1):83-90. doi: 10.1097/00000539-199901000-00016. PMID 9895071
- [Background] Myles PS, Weitkamp B, Jones K, Melick J, Hensen S. Validity and reliability of a postoperative quality of recovery score: the QoR-40. Br J Anaesth. 2000 Jan;84(1):11-5. doi: 10.1093/oxfordjournals.bja.a013366. PMID 10740540
- [Background] Insall JN, Dorr LD, Scott RD, Scott WN. Rationale of the Knee Society clinical rating system. Clin Orthop Relat Res. 1989 Nov;(248):13-4. PMID 2805470
- [Background] Melvin JS, Stryker LS, Sierra RJ. Tranexamic Acid in Hip and Knee Arthroplasty. J Am Acad Orthop Surg. 2015 Dec;23(12):732-40. doi: 10.5435/JAAOS-D-14-00223. Epub 2015 Oct 22. PMID 26493971
- [Derived] Heller S, Shemesh S, Rukinglaz O, Cohen N, Velkes S, Fein S. Efficacy of single-shot adductor canal block before Versus after primary total knee arthroplasty - Does timing make a difference? A randomized controlled trial. J Orthop Surg (Hong Kong). 2022 Sep-Dec;30(3):10225536221132050. doi: 10.1177/10225536221132050. PMID 36189733